CLINICAL TRIAL: NCT00281671
Title: Pilot Study of the Effects of Nesiritide on Hemodynamics and Urine Output Following Cardiopulmonary Bypass in Infants
Brief Title: Nesiritide Use Following Cardiac Surgery in Infants
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow patient enrollment.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, John M Costello, Attending Physician, Department of Cardiology, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-12-160
Record Dates: First submitted 2006-01-23; First posted 2006-01-25 (Estimated); Results first posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2018-05

CONDITIONS: Heart Defects, Congenital; Cardiopulmonary Bypass
Keywords: Nesiritide; Natriuretic Peptide, Brain; Heart Defects, Congenital; Cardiopulmonary Bypass; Diuretics
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Natriuretic Peptide, Brain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): In this crossover pilot study, patients are randomly assigned to receive either nesiritide or placebo infusion for 10 hours, followed by a two hour washout period, and then the other study drug for 10 hours.
  Interventions: Drug: Placebo
- Nesiritide (Experimental): In this crossover pilot study, patients are randomly assigned to receive either nesiritide or placebo infusion for 10 hours, followed by a two hour washout period, and then the other study drug for 10 hours.
  Interventions: Drug: nesiritide

INTERVENTIONS:
Drug: nesiritide — nesiritide 0.015 mcg/kg/hour x 10 hours
  Other Names: Natrecor
  Arms: Nesiritide
Drug: Placebo — 0.9% sodium chloride infusion
  Other Names: 0.9% sodium chloride infusion
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of nesiritide on urine output and hemodynamics following cardiopulmonary bypass in infants. Safety and pharmacokinetic data will also be obtained.

DETAILED DESCRIPTION:
Nesiritide, a recombinant human B-type natriuretic peptide, has vasodilatory, lusitropic and diuretic properties in healthy humans, and improves hemodynamics and symptoms in adults with decompensated congestive heart failure. Several retrospective case series suggest that nesiritide has beneficial effects on hemodynamics and urine output in adults and children following cardiac surgery.

The purpose of this prospective, randomized, double-blind, crossover study is to evaluate the effects of a continuous infusion of nesiritide on postoperative hemodynamics and urine output in infants with congenital heart disease who undergo cardiac surgery requiring cardiopulmonary bypass (CPB). Patients less than 1 year of age following cardiac surgery will be eligible for the study if they have received two conventional diuretics (furosemide and chlorothiazide) for at least 12 hours, yet are not effectively achieving a negative fluid balance, thus prohibiting sternal closure or tracheal extubation. Patients will be randomized to receive either a 10-hour infusion of nesiritide, a two hour washout period, followed by a 10-hour infusion of placebo, or this study drug sequence in reverse order. During the 24-hour study period, serial cardiac output measurements and BNP levels will be obtained, vital signs and intracardiac filling pressures will be recorded, and urine output will be measured.

ELIGIBILITY:
Inclusion Criteria:

* > 48 hours after cardiac surgery requiring cardiopulmonary bypass
* < 1 year of age
* Receiving chlorothiazide and furosemide for > 12 hours
* Urine output < 4 cc/kg/hour, or fluid intake > output for 2 consecutive days
* Receiving mechanical ventilation
* Presence of body wall edema on CXR, defined as a radiologic index of > 2
* Plan for > 24 hrs further diuresis before chest closure or extubation

Exclusion Criteria:

* Age > 365 days at the time of enrollment
* Corrected estimated gestational age < 35 weeks at the time of enrollment
* Serum creatinine > 2.0 mg/dL at the time of enrollment
* Significant hemodynamic instability at the time of enrollment
* Lack of dedicated intravenous access for nesiritide infusion
* Lack of arterial line for continuous blood pressure monitoring
* Lack of a Foley catheter for continuous urine collection
* Enrollment in another research study such that the outcomes of either study may be confounded by participation in this study, or such that the amount of blood drawn for research purposes becomes excessive.

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2006-04-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John M Costello, MD, Principal Investigator — Department of Cardiology, Children's Hospital Boston
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Email PI for data requests.

REFERENCES:
- [Background] Costello JM, Backer CL, Checchia PA, Mavroudis C, Seipelt RG, Goodman DM. Effect of cardiopulmonary bypass and surgical intervention on the natriuretic hormone system in children. J Thorac Cardiovasc Surg. 2005 Sep;130(3):822-9. doi: 10.1016/j.jtcvs.2005.03.008. PMID 16153935
- [Background] Costello JM, Backer CL, Checchia PA, Mavroudis C, Seipelt RG, Goodman DM. Alterations in the natriuretic hormone system related to cardiopulmonary bypass in infants with congestive heart failure. Pediatr Cardiol. 2004 Jul-Aug;25(4):347-53. doi: 10.1007/s00246-003-0512-5. PMID 14735254
- [Background] Mahle WT, Cuadrado AR, Kirshbom PM, Kanter KR, Simsic JM. Nesiritide in infants and children with congestive heart failure. Pediatr Crit Care Med. 2005 Sep;6(5):543-6. doi: 10.1097/01.pcc.0000164634.58297.9a. PMID 16148814
- [Background] Simsic JM, Reddy VS, Kanter KR, Kirshbom PM, Forbess JM. Use of nesiritide (human B-type natriuretic peptide) in infants following cardiac surgery. Pediatr Cardiol. 2004 Nov-Dec;25(6):668-70. doi: 10.1007/s00246-003-0680-3. PMID 14994182

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment: April 2006- June 2007.
  Location: Cardiac ICU in a large children's hospital.
Groups:
- Nesiritide First, Then Placebo: Patients assigned to this arm received nesiritide 0.015 mcg/kg/hour for 10 hours, followed by a two hour washout period, and then a placebo infusion (0.9 normal saline) for 10 hours
- Placebo First, Then Nesiritide: Patients assigned to this arm received a placebo infusion (0.9 normal saline) for 10 hours, followed by a two hour washout period, and then nesiritide 0.015 mcg/kg/hour for 10 hours
Period: Overall Study
Arm/Group | Nesiritide First, Then Placebo | Placebo First, Then Nesiritide
Started | 5 | 4
Completed | 5 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Because all participants were randomized to receive all interventions, baseline measurements are combined rather that reported by Arm/Group.
Arm/Group | All Study Participants
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: days] | 6 [4 to 103]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants] — Northeast United States
  participants
    United States | 9
Weight [Median (Full Range); unit: Kg] | 3.5 [2.5 to 4.9]
Prematurity [Count of Participants; unit: Participants] | 2

OUTCOME MEASURES:

1. Primary Outcome: Urine Output
Description: Urine output measured in cc/kg/hour during the last 5 hours of the study drug infusion
Time Frame: 5 hours
Measure: Median (Full Range); unit: cc/kg/hr
Groups:
- Placebo: In this crossover pilot study, patients were randomly assigned to receive either nesiritide 0.015 mcg/kg/min or placebo IV infusion for 10 hours, followed by a two hour washout period, and then the other study drug for 10 hours.
  For this arm, the data reflect the urine output during the last 5 hours of the 0.9 normal saline placebo infusion for all 9 patients.
- Nesiritide: In this crossover pilot study, patients are randomly assigned to receive either nesiritide 0.015 mcg/kg/min or placebo IV infusion for 10 hours, followed by a two hour washout period, and then the other study drug for 10 hours.
  For this arm, the data reflect the urine output during the last 5 hours of the nesiritide 0.015 mcg/kg/hour infusion for all 9 patients.
Arm/Group | Placebo | Nesiritide
Number analyzed (Participants) | 9 | 9
cc/kg/hr | 2.9 [1.1 to 7.1] | 3.1 [0.6 to 6.4]

2. Secondary Outcome: Number of Participants With Hypotension and Bradycardia
Description: Hypotension (mean arterial blood pressure < 40 mmHg for > 30 minutes) that is refractory to volume administration, increased inotropic/vasopressor support, and weaning of other vasodilators (e.g., milrinone) or sedatives
  Bradycardia, defined as 1) a decrease in heart rate of more than 30 beats/minute from baseline following the initiation of study drug infusion that 2) results in new requirement for temporary atrial pacing or other treatment specifically to increase heart rate and 3) is not readily explainable by other conditions.
Time Frame: 48 hours
Measure: Count of Participants; unit: Participants
Groups:
- Nesiritide: In this crossover pilot study, patients are randomly assigned to receive either nesiritide or placebo infusion for 10 hours, followed by a two hour washout period, and then the other study drug for 10 hours.
  For this arm, the data reflect the urine output during the last 5 hours of the nesiritide 0.015 mcg/kg/hour infusion for all 9 patients.
Arm/Group | Placebo | Nesiritide
Number analyzed (Participants) | 9 | 9
Participants
  hypotension | 0 | 0
  bradycardia | 0 | 0

3. Secondary Outcome: Urine Output
Time Frame: 10 hours
Measure: Median (Full Range); unit: cc/kg/hr
Groups:
- Placebo; Nesiritide: In this crossover pilot study, patients are randomly assigned to receive either nesiritide 0.015 mcg/kg/min or placebo IV infusion for 10 hours, followed by a two hour washout period, and then the other study drug for 10 hours.
  nesiritide: nesiritide 0.015 mcg/kg/hour x 10 hours
Arm/Group | Placebo | Nesiritide
Number analyzed (Participants) | 9 | 9
cc/kg/hr | 3.4 [1.1 to 6.0] | 4.2 [1.3 to 5.7]

4. Secondary Outcome: Cardiac Index
Description: Cardiac index is based on the cardiac output, which is the amount of blood the left ventricle ejects into the systemic circulation in one minute, measured in liters per minute (l/min). Cardiac output is indexed to a patient's body size by dividing by the body surface area (m^2) to yield the cardiac index. Cardiac index was calculated in patients with an SVC catheter (previously placed for clinical indications) using the Fick principle using measured oxygen consumption (VO2), hemoglobin levels, and the difference between arterial and superior vena cava oxygen saturation. Oxygen consumption was measured using a real-time gas exchange technique with the Deltatrack II gas sensor.
Time Frame: Baseline (hour 0) and 6 hours after onset of study drug infusion
Population: Cardiac index was only able to be measured for 4 of the 9 subjects enrolled in the trial.
Measure: Median (Full Range); unit: L/min/m^2
Arm/Group | Placebo | Nesiritide
Number analyzed (Participants) | 4 | 4
L/min/m^2
  baseline | 1.83 [0.95 to 3.61] | 1.90 [1.50 to 3.26]
  6 hours after onset of drug infusion | 1.95 [1.40 to 5.80] | 2.15 [1.42 to 3.67]

ADVERSE EVENTS:
Time Frame: Initiation of study interventions until 48 hours after the study drug infusions ended.
Groups:
- Nesiritide: Patients received nesiritide 0.015 mcg/kg/hour for 10 hours
- Placebo: Patients assigned to this arm received a placebo infusion (0.9 normal saline) for 10 hours
Arm/Group | Nesiritide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No